CLINICAL TRIAL: NCT07349043
Title: A Prospective, Safety, and Efficacy Clinical Trial of Pressurized Intraperitoneal Aerosol Therapy for Peritoneal Metastasis of Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1055
Record Dates: First submitted 2025-12-04; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Peritoneal Metastasis; CRC (Colorectal Cancer)
Keywords: peritoneal metastasis; CRC; PIPAC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The MTD of PIPAC combined with mitomycin (MMS) in the treatment of CRCPM (Experimental): This trial is a prospective study, and the subjects are patients diagnosed with peritoneal metastasis of colorectal cancer.
  Mitomycin-PIPAC group: The patients were treated with mitomycin (increasing dose: 5mg/m2, 10mg/m2, 15mg/m2, 20mg/m2) + 0.9% saline 50 mL by pressurized intraperitoneal aerosol chemotherapy.
  PIPAC frequency: 1 time/4-6W, continuous treatment for 3 courses (if the subject is unable to undergo the second or third PIPAC, the investigator needs to record the reason).
  3.6.2 Surgical plan The principle of mesenteric resection and tumor-free operation should be followed in tumor reduction surgery.
  3.6.3 Systemic chemotherapy regimen The chemotherapy regimen is determined by clinicians based on pathological staging, molecular typing, risk factors, and in accordance with the guidelines of the NCCN and CSCO.
  Interventions: Drug: Mitomycin-PIPAC
- The MTD of PIPAC combined with raloxifene (RTX) in the treatment of CRCPM (Experimental): This trial is a prospective study, and the subjects are patients diagnosed with peritoneal metastasis of colorectal cancer.
  Raltitrexed-PIPAC group: Raltitrexed (dose escalation: 1mg/m2, 1.5mg/m2, 2mg/m2, 2.5mg/m2, 3mg/m2) + 0.9% saline 50 mL for pressurized intraperitoneal aerosol chemotherapy.
  PIPAC frequency: 1 time/4-6W, continuous treatment for 3 courses (if the subject is unable to undergo the second or third PIPAC, the investigator needs to record the reason).
  3.6.2 Surgical plan The principle of mesenteric resection and tumor-free operation should be followed in tumor reduction surgery.
  3.6.3 Systemic chemotherapy regimen The chemotherapy regimen is determined by clinicians based on pathological staging, molecular typing, risk factors, and in accordance with the guidelines of the NCCN and CSCO.
  Interventions: Drug: Raltitrexed-PIPAC

INTERVENTIONS:
Drug: Mitomycin-PIPAC — Mitomycin-PIPAC group: The patients were treated with mitomycin (increasing dose: 5mg/m2, 10mg/m2, 15mg/m2, 20mg/m2) + 0.9% saline 50 mL by pressurized intraperitoneal aerosol chemotherapy.
  Arms: The MTD of PIPAC combined with mitomycin (MMS) in the treatment of CRCPM
Drug: Raltitrexed-PIPAC — Raltitrexed-PIPAC group: Raltitrexed (dose escalation: 1mg/m2, 1.5mg/m2, 2mg/m2, 2.5mg/m2, 3mg/m2) + 0.9% saline 50 mL for pressurized intraperitoneal aerosol chemotherapy.
  Arms: The MTD of PIPAC combined with raloxifene (RTX) in the treatment of CRCPM

SUMMARY:
For colorectal cancer with peritoneal metastasis, the current first-line standard treatment offers very limited benefits and short survival. Therefore, it is necessary to seek new treatment strategies to improve the prognosis and survival of such patients. Based on previous basic research and early clinical research results, the strategy of PIPAC combined with MMC or RTX provides a feasible solution that can benefit patients with advanced colorectal cancer and peritoneal metastasis undergoing first-line treatment. This study aims to evaluate the effectiveness of PIPAC combined with MMC or RTX as first-line treatment for patients with colorectal cancer and peritoneal metastasis, while ensuring that patients receive standard first-line treatment. (The main purpose of the proposed Phase I trial is to determine the MTD of PIPAC combined with MMC or RTX and evaluate the safety of combining it with systemic chemotherapy for patients with colorectal cancer and peritoneal metastasis.)

DETAILED DESCRIPTION:
1. Research background Colorectal cancer (CRC) is one of the most common malignant tumors. Globally, approximately 1 million new cases of colorectal cancer occur each year, and about 500,000 people die from the disease annually. With the improvement of living standards and changes in lifestyle habits, the incidence rate of colorectal cancer is gradually increasing, posing a serious threat to human life. To prevent the occurrence of peritoneal metastasis, based on previous basic research and early clinical research results, the strategy of PIPAC combined with MMC or raltitrexed provides a feasible approach that can benefit patients with advanced colorectal cancer who undergo first-line treatment for peritoneal metastasis.
2. Research purpose To evaluate the safety and determine the maximum tolerated dose (MTD) of pressurized intraperitoneal aerosol chemotherapy combined with mitomycin or raltitrexed in patients with colorectal cancer and peritoneal metastasis.

II. Specific Procedures and Processes

1. Treatment method This trial is a prospective study, and the subjects are patients diagnosed with peritoneal metastasis of colorectal cancer.

   Mitomycin-PIPAC group: Mitomycin (increasing doses: 5mg/m2, 10mg/m2, 15mg/m2, 20mg/m2) + 0.9% saline 50 mL was administered via intraperitoneal aerosol chemotherapy under pressure.

   Raltitrexed-PIPAC group: Raltitrexed (dose escalation: 1mg/m2, 1.5mg/m2, 2mg/m2, 2.5mg/m2, 3mg/m2) + 0.9% saline 50 mL for pressurized intraperitoneal aerosol chemotherapy.

   PIPAC frequency: 1 time/4-6W, continuous treatment for 3 courses (if the subject is unable to undergo the second or third PIPAC, the investigator needs to record the reason).

   Equipment: Pressure Intraperitoneal Aerosol Chemotherapy (PIPAC) equipment includes an endoscope pulse irrigation device and its supporting instruments, mainly including a display screen, an infusion rack, a liquid sensor, a high-pressure peristaltic pump, and the main structure of the machine; supporting instruments include: 10 mm atomizing nozzle, high-pressure infusion tube, infusion tube puncture head, and 10/12 mm trocar puncture device (2).

   Surgical plan The principle of mesenteric resection and tumor-free operation should be followed in tumor reduction surgery.

   systemic chemotherapy regimen The chemotherapy regimen is determined by the clinician based on pathological staging, molecular typing, risk factors, and in accordance with the NCCN and CSCO guidelines.
2. Visit and follow-up Patients came to the hospital for follow-up visits according to the requirements of the research protocol and continued until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peritoneal metastatic adenocarcinoma of colorectal origin, confirmed by histopathology, and without metastasis to other sites.
2. No gender limitation, aged 18 to 75 years old;
3. ECOG score ≤2;
4. Subjects without other malignant diseases;
5. Subjects without laparoscopic surgery contraindications;
6. Expected survival period > 6 months;
7. Able to comprehend and sign the informed consent form;
8. The function of important organs should meet the following requirements; The absolute neutrophil count (ANC) is ≥1.5×10^9/L; Platelets ≥ 100×10^9/L; Hemoglobin ≥8.0g/dl (Note: It is acceptable to achieve hemoglobin ≥8.0g/dl through blood transfusion or other interventions); serum albumin ≥2.8g/dL; Bilirubin ≤1.5 times ULN, ALT and AST ≤1.5 times ULN; if there is liver metastasis, ALT and AST ≤5 times ULN; Creatinine clearance rate ≥50mL/min

Exclusion Criteria:

1. Subjects with gastrointestinal obstruction;
2. Subjects who rely entirely on parenteral nutrition;
3. Subjects with decompensated ascites;
4. Subjects with severe abdominal infection (peritonitis);
5. Subjects with extensive abdominal adhesion;
6. Subjects who underwent both tumor reduction surgery and gastrointestinal resection and reconstruction simultaneously;
7. Subjects with portal vein thrombosis;
8. Patients with severe or uncontrolled medical conditions and infections (including atrial fibrillation, angina pectoris, heart failure, ejection fraction less than 50%, refractory hypertension, etc.);
9. Previously allergic to chemotherapy drugs;
10. Individuals with severe heart and lung, liver and kidney, blood system, or mental illnesses, as well as those who abuse drugs;
11. Pregnant or lactating women;
12. Patients who have participated in or are currently participating in other clinical trials within 3 months;
13. Other situations where the researchers believe that the patient is not suitable to participate in this trial;
14. Previously had a history of neurological or psychiatric disorders that would affect study informed consent or follow-up evaluation, such as severe depression or dementia;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | the first 4 weeks
  The number and severity of toxicities observed during treatment, as well as their relation to the dose level of MMS or RTX administered via PIPAC.
Maximum Tolerated Dose (MTD) | 4 weeks
  MTD will be determined based on the highest dose administered where <33% of patients experience DLTs, or by dose-escalation schemes according to standard practices.
Adverse Events (AEs) | up to 12 months
  Monitoring and documenting all adverse events (e.g., nausea, fatigue, pain, hematological effects) following each dose escalation.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 48h
  To measure the highest plasma concentration of mitomycin (MMS) or raltitrexed (RTX) after PIPAC administration.
Objective Response Rate (ORR) | up to 12 months
  Measured using imaging techniques and clinical assessment to determine the proportion of patients who achieve complete or partial response.
Progression-Free Survival (PFS) | up to 12 months
  Time from treatment initiation to disease progression or death from any cause.
Overall Survival (OS) | up to 12 months
  Time from treatment initiation to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine 88 Jiefang Road Hangzhou, Zhejiang 310009, China, Hangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns and the sensitive nature of the health information collected, which cannot be sufficiently de-identified for sharing.